CLINICAL TRIAL: NCT01202695
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation Study Evaluating Pharmacokinetics and Safety of a Human Monoclonal Antibody (AVP-21D9) in Normal Healthy Volunteers
Brief Title: Safety and Pharmacokinetics Study of Human Monoclonal Antibody (AVP-21D9)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EBS.AVP.001; DMID 09-0008 (Other Grant/Funding Number: HHSN272200800040C)
Record Dates: First submitted 2010-09-13; First posted 2010-09-16 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Anthrax
MeSH Terms: conditions — Anthrax | interventions — AVP-21D9

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AVP-21D9 (Experimental)
  Interventions: Drug: AVP-21D9
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVP-21D9 — intravenously, single dose
  Arms: AVP-21D9
Drug: Placebo — Placebo comparator
  Other Names: Placebo comparator
  Arms: Placebo

SUMMARY:
Primary:

• To compare the safety profile of a single intravenous administration of AVP-21D9 as compared with Placebo

Secondary:

* To evaluate the pharmacokinetics (PK) of a single intravenous administration of AVP-21D9
* To evaluate the immunogenicity of AVP-21D9

DETAILED DESCRIPTION:
This is a sequential, dose-escalating healthy volunteer study of the safety and pharmacokinetics of intravenously-infused AVP-21D9.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy volunteers, between 18 and 45 years of age
* Normal laboratory (blood test) results

Key Exclusion Criteria:

* Prior immunization with anthrax vaccine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety assessments | 90 days following infusion
  Safety will be assessed by collecting data (physical exams, adverse event reporting, lab testing/analysis) and concomitant medications at each visit from pre-infusion period through post-infusion day 90 or the early withdrawl visit, if applicable.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) analysis | 90 days following infusion
  PK parameters will be determined for a single intravenous administration of AVP-21D9 as measured by an immunoassay for AVP-21D9.
Immunogenicity analysis | From day 1 up to day 90 following infusion
  Immunogenicity will be measured by blood testing/analysis on anti-AVP-21D9 antibody generation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hopkins, MD, Study Director — Emergent BioSolutions
Locations (1):
- ICON Development Solutions, San Antonio, Texas, United States

REFERENCES:
- [Derived] Malkevich NV, Hopkins RJ, Bernton E, Meister GT, Vela EM, Atiee G, Johnson V, Nabors GS, Aimes RT, Ionin B, Skiadopoulos MH. Efficacy and safety of AVP-21D9, an anthrax monoclonal antibody, in animal models and humans. Antimicrob Agents Chemother. 2014 Jul;58(7):3618-25. doi: 10.1128/AAC.02295-13. Epub 2014 Apr 14. PMID 24733473